CLINICAL TRIAL: NCT03811496
Title: Biomarker Analysis for Parkinson's Disease in Subjects With Glucocerebrosidase Mutations
Brief Title: Biomarker Analysis for GBA Associated Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-LDRTC-01
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease; Gaucher Disease
Keywords: Parkinson disease; Gaucher disease; GBA gene; alpha-synuclein
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GD-PD: Patients and carriers of Gaucher disease with confirmed mutations in GBA gene who have developed Parkinson's disease symptoms
- GD-nonPD: Patients with Gaucher disease but no known Parkinson's symptoms
- nonGD-nonPD: Non-Gaucher disease/healthy controls

SUMMARY:
The primary aim of the study is to conclusively demonstrate the possibility of using the following molecules, α-Synuclein, LRRK2 and Parkin individually or in combination as biomarkers for Parkinson's disease (PD) progression in patients/ carriers of Gaucher disease (GD). All the assays will be performed only using peripheral blood, thus the identification of a peripheral marker that can be used in both diagnosis and prognosis of the disease and symptom severity would lead to a fast, efficient and reliable assay that can be performed on an easily accessible tissue type outside of the brain. It is now known that patients with GD, even carriers with one mutated GBA gene (OMIM 606463) are at a higher risk for developing PD, and at an earlier age. In an attempt to assess whether GBA alterations would also impact α-Synuclein and Parkin metabolism in humans, the expression at both molecular and protein level in the peripheral blood mononuclear cells (PBMCs) will be investigated.

DETAILED DESCRIPTION:
The GBA (OMIM 606463) gene codes for beta-glucocerebrosidase, a lysosomal enzyme. Disease causing mutations in both alleles of GBA gene cause Gaucher disease (GD) while mutations in one allele lead to Gaucher carrier status. It has been shown recently that patients with GD, even carriers with one mutated GBA gene are at a higher risk for developing Parkinson disease (PD), and at an earlier age, and that the GBA mutations comprise the primary genetic risk factor in the development of PD and other forms of parkinsonism. However, there are no biomarkers to determine the diagnosis of PD, especially in the early and minimally symptomatic or asymptomatic stage. The progression of PD in subjects with a mutation in the GBA gene can currently not be determined. In some cellular and animal models, glucocerebrosidase alterations were shown to impact the metabolism of other proteins implicated in PD pathology. α-Synuclein and Parkin, encoded by SNCA and PARK2 respectively, are implicated in rare genetic forms of parkinsonism. α-Synuclein aggregates are seen in cells of the central and peripheral nervous system and is considered to be the pathological culprit in PD. Mutated glucocerebrosidase has been shown to be present in α-Synuclein aggregates in postmortem brain samples from individuals with GBA mutations and PD. α-Synuclein in addition, is shown to affect the solubility of Parkin in the cells. As an attempt to assess whether GBA alterations would also impact α-Synuclein and Parkin metabolism in humans in easily accessible cell types outside the brain, the expression at both molecular and protein level will be investigated in the peripheral blood mononuclear cells (PBMCs). The study includes three cohorts: 1) Patients and carriers of Gaucher disease with confirmed disease causing mutations in GBA gene who have developed Parkinson's disease symptoms (GD-PD), 2) Patients and carriers of Gaucher disease with no known Parkinson's symptoms (GD-nonPD) and 3) Non-Gaucher disease/healthy controls (HC). PBMCs extracted from 3-5 ml peripheral blood will be used for intracellular staining for α-Synuclein, LRRK2 and Parkin and then acquired on Flow cytometer (BD accuri). Lymphocytes and monocytes will be analyzed for α-Synuclein, LRRK2 and Parkin expression. PBMCs will also be used for RNA extraction and subsequent molecular analysis using qPCR. Since the assay utilizes an easily accessible tissue type i.e., peripheral blood and requires a very small amount (2-3 ml), this assay could be developed as a potential biomarker for diagnosis and a disease progression indicator for Parkinson disease in subjects with GBA gene mutations.

ELIGIBILITY:
Inclusion Criteria:

The study will include

1. adult subjects age 21 or older with Gaucher disease with and without parkinsonism and individuals from families with a Gaucher proband and a history of parkinsonism.
2. Controls will include unaffected siblings of patients with Gaucher disease and subjects with sporadic PD, without glucocerebrosidase mutations, and healthy volunteers who do not have a family history of parkinsonism or Gaucher disease.

Exclusion Criteria:

Subjects excluded from the study include those who:

1. present with severe cognitive deficits impairing decision making
2. are unable to or for whom it is medically unsafe to withdraw from their current medications, such as subjects on SSRI s and other psychoactive drugs. The subjects on SSRIs may be included in the study only with an approval from the prescribing physician to discontinue their medications temporarily for the study.
3. are pregnant or nursing. All women of child bearing potential will undergo a pregnancy test.
4. have a history of neurologic conditions such as stroke or any focal brain lesion that may result in parkinonian manifestations. Individuals with such MRI findings will be excluded from the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study will include three cohorts:
  1. Patients and carriers of Gaucher disease with confirmed mutations in GBA gene who have developed Parkinson's disease symptoms (GD-PD),
  2. Patients with Gaucher disease but no known Parkinson's symptoms (GD-nonPD) and
  3. Non-Gaucher disease/healthy controls (nonGD-nonPD). All participants will be recruited after obtaining informed consent using IRB (Independent Review Board) approved informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Gene expression levels of SNCA | 18 months
  Gene expression levels relative to internal reference genes will be compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression of SNCA.
Gene expression levels of LRRK2 | 18 months
  Gene expression levels relative to internal reference genes will be compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression of LRRK2.
Gene expression levels of Parkin | 18 months
  Gene expression levels relative to internal reference genes will be compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression of Parkin.
Protein expression levels of alpha-synuclein | 18 months
  Protein expression levels of alpha-synuclein will be analyzed using flow cytometry and compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression.
Protein expression levels of LRRK2 | 18 months
  Protein expression levels of LRRK2 will be analyzed using flow cytometry and compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression.
Protein expression levels of Parkin | 18 months
  Protein expression levels of Parkin will be analyzed using flow cytometry and compared between the individual subjects as well as grouped analysis to identify a specific pattern in alterations in level of expression.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — LDRTC; Renuka Limgala, PhD, Principal Investigator — LDRTC
Locations (1):
- LDRTC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Institute website for more details — http://www.ldrtc.org